CLINICAL TRIAL: NCT04244032
Title: Cognitive Enhancement Through Computerized Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment barriers
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB201901330; K01AA026893 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder
Keywords: Cognitive Training; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Working Memory Training (WM) (Experimental): Participants complete training in a working memory task designed to utilize individually-adapted difficulty levels.
  Interventions: Behavioral: Working Memory Training
- Inhibitory Control Training (IC) (Experimental): Participants complete training in an inhibitory control task designed to utilize individually-adapted difficulty levels.
  Interventions: Behavioral: Inhibitory Control Training
- Bias Modification Training (BM) (Active Comparator): Participants complete training in an active comparator task designed to weaken approach responses to alcohol-associated cues.
  Interventions: Behavioral: Bias Modification Training
- Non-Trained control (NTC) (No Intervention): No active intervention is delivered beyond typical care.

INTERVENTIONS:
Behavioral: Working Memory Training — Participants complete up to 12 sessions of computerized training (30-45 min each) in a working memory task designed to utilize individually-adapted difficulty levels.
  Arms: Working Memory Training (WM)
Behavioral: Inhibitory Control Training — Participants complete up to 12 sessions of computerized training (30-45 min each) in an inhibitory control task designed to utilize individually-adapted difficulty levels.
  Arms: Inhibitory Control Training (IC)
Behavioral: Bias Modification Training — Participants complete up to 12 sessions of computerized training (30-45 min each) in a bias modification task designed to utilize individually-adapted difficulty levels.
  Arms: Bias Modification Training (BM)

SUMMARY:
Alcohol use disorder is characterized by widespread neurocognitive impairments, however despite substantial advances in the intervention and treatment of alcohol use disorders, exceptionally few studies have been directed to improving these deficits. This project leverages computerized cognitive training, applied as an adjunct to inpatient treatment, to enhance neurocognitive recovery. This project informs public health and future intervention efforts by interrogating factors critical to intervention efficacy and clarifying relationships between neurocognitive recovery and treatment outcomes, including post-discharge alcohol consumption.

DETAILED DESCRIPTION:
Programmatic investigation of neurocognitive functioning in alcohol use disorder (AUD) has revealed widespread and sustained impairments. Despite conceptual relevance to treatment efficacy, few AUD interventions have been directed to the remediation of these impairments. This project is responsive to this gap. It will answer critical questions regarding the potential of cognitive training (CT), applied as an adjunct to inpatient treatment, to improve cognitive recovery and post-discharge functional outcomes in AUD.

The current project will investigate the efficacy of two experimental cognitive training interventions in a sample of inpatients in treatment for AUD. While the effectiveness of CT to enhance function is supported by diverse literatures, it remains largely unexamined in AUD. The current project will interrogate the degree to which cognitive training interventions can "transfer" cognitive gains to untrained tasks/domains, and improve overall executive functioning. It will apply conceptual models from the CT and alcohol literatures to identify factors associated with CT efficacy. The impact of cognitive training on functional outcomes, including post-discharge drinking, will be investigated. Finally, relationships between cognitive recovery during treatment and post-discharge adaptation will be examined. Thus, the current work will be of substantial import to public health, alcohol science, and will inform future intervention efforts.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 10 years of education
* Meet DSM-5 criteria for alcohol use disorder

Exclusion Criteria:

* Medical histories confounding interpretation regarding change in neuropsychological functioning (e.g., stroke)
* Meet DSM-5 criteria for current/unremitted psychotic, panic, or bipolar disorders

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Working Memory | Baseline and up to 3 weeks
  Performance on neuropsychological measures indexing working memory capacity. Score range: 0-100 (scores <40 are poor [0-16th percentile]; scores >60 are good [84th-100th percentile]).
Inhibitory Control | Baseline and up to 3 weeks
  Performance on neuropsychological measures indexing inhibitory control capacity. Score range: 0-100 (scores <40 are poor [0-16th percentile]; scores >60 are good [84th-100th percentile]).
General Executive Function | Baseline and up to 3 weeks
  Performance on neuropsychological measures indexing general executive functioning. Score range: 0-100 (scores <40 are poor [0-16th percentile]; scores >60 are good [84th-100th percentile]).

CONTACTS AND LOCATIONS:
Overall Officials: Ben Lewis, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No